CLINICAL TRIAL: NCT02711670
Title: Night-time Use of Thiazide Diuretics for Improved Reduction in Stone Risk in Stone Formers With Elevated Urine Calcium
Brief Title: Night Time Use of Thiazide Diuretics for Improved Reduction in Stone Risk in Stone Formers With Elevated Urine Calcium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, David S. Goldfarb, M.D., PI, VA New York Harbor Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01417
Record Dates: First submitted 2015-02-04; First posted 2016-03-17 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Kidney Stones
Keywords: nephrolithiasis; calcium stones; kidney stones; hypercalciuria; thiazide
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Hypercalciuria | interventions — Chlorthalidone; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thiazide (Experimental): Stone formers History of calcium containing kidney stones, hypercalciuria on previous urine tests, no kidney disease, not pregnant/lactating
  Interventions: Drug: chlorthalidone; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: chlorthalidone
Drug: Hydrochlorothiazide

SUMMARY:
Thiazide diuretics will be more effective in lowering urine calcium excretion if taken at night as compared to the daytime. It will therefore be more effective in reducing kidney stone recurrence in nephrolithiasis patients with elevated urine calcium who are known to have increased risk of kidney stones at night time.

DETAILED DESCRIPTION:
The study will be divided into three phases for every single patient, investigators will study 15-20 stone formers who have previously documented elevated urine calcium excretion, with a plan to measure their urine chemistries at baseline (if they currently use thiazide diuretics, they will come off of their respective thiazide for a 7-day washout period). Investigators will ask them to collect urine samples in two 12-hour intervals: on awakening, the 1st sample starts to before supper; 2nd sample begins after dinner and extends overnight with fasting after dinner, These measurements will be used as controls. Then patients will be started back on diuretics (25mg of chlorthalidone for the primary study; pending the results this may be repeated with 25mg of hydrochlorothiazide as a second substudy) which they will take in the daytime; after a 6-day acclimation period, two 12-hour urine samples will be collected as in the washout period. For the third study period, the patients will then begin taking the thiazide after dinner. After a 6-day acclimation period, the third set of urine collections will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent calcium kidney stones (at least 2 episodes) and either a higher urine calcium excretion (urine Ca >200 mg/d or > 4 mg/kg body weight) or,
* In patients who currently take a thiazide diuretic, a history of elevated urine calcium prior to medication use;
* Also capable of signing consent and doing 24-hour urine collections repeatedly.

Exclusion Criteria:

* Patients with primary hyperparathyroidism, renal tubular acidosis, chronic kidney disease (serum creatinine > 1.5 mg/dl), inflammatory bowel disease, gout,
* Patients taking thiazides with a history of hypertension,
* Patients with baseline systolic blood pressure less than 110mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in excretion and supersaturation of urine calcium oxalate / phosphate | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — New York Harbor VA Medical Center
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States